CLINICAL TRIAL: NCT00491010
Title: Maximum Targeted Ablation of Atrial Flutter
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-06-153; 12266
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Atrial Flutter
Keywords: atrial flutter; ablation; voltage targeted
MeSH Terms: conditions — Atrial Flutter | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: radiofrequency catheter ablation

SUMMARY:
Patients undergoing atrial flutter ablation will be randomized to either the standard ablation approach or voltage targeted approach. Patients will be followed for one year to assess outcome of the ablation technique

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing TV-IVC isthmus ablatin for atrial flutter

Exclusion Criteria:

* atypical atrial flutter
* <18 years old any atrial surgery or pacemaker refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-07; Study Completion 2008-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Allan c Skanes, MD, Principal Investigator — University of Western Ontario, London Health Sciences Center
Locations (1):
- London Health Sciences Center, London, Ontario, Canada